CLINICAL TRIAL: NCT01395212
Title: Long-term Follow-up of Patients With Ischemic Heart Disease Treated With Combined Delivery of Autologous Bone-marrow Mononuclear Cells: 5-year Clinical Outcome of the MYSTAR Study
Brief Title: MYSTAR-5-YEAR: Long-term Follow-up of Patients With Ischemic Heart Disease Treated With Cell Therapy
Acronym: MYSTAR-5-YEAR
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Mariann Gyongyosi, Prof. Dr., Medical University of Vienna
Other Study IDs: MUW
Record Dates: First submitted 2011-07-14; First posted 2011-07-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Acute Myocardial Infarction
Keywords: Cell-based cardiac regenerative therapy; Intramyocardial injections; NOGA procedure; Acute myocardial infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac stem cell therapy 5 years ago

SUMMARY:
The MYSTAR-5-YEAR study controls the patients 5 years after treatment with combined (intramyocardial and intracoronary) delivery of autologous BM-MNCs.

The clinical endpoint of this prospective non-randomized observational study is the MACCE, defined as major adverse cardiac and cerebrovascular events. Patients will be investigated by echocardiography, SPECT and MRI. 2D (NOGA-guided SPECT) and 3D (NOGA-guided MRI) imaging will refine the evaluation with more exact analysis of the intramyocardial injected areas (ROI).

DETAILED DESCRIPTION:
Background: Based on the available long-term results of cardiac stem cell therapies, it seems, that it offers short-term moderate benefits, but the long-term outcome is still matter of debate. In 2008, the Austrian arm of the MYSTAR study (a prospective multi-center single-blind trial) including patients with recent AMI and treated with combined (intramyocardial and intracoronary) delivery of autologous BM-MNCs has been completed with 1-year FUP. The MYSTAR results showed moderate but significant improvement in infarct size and LV function similar to other trials, and confirmed safety, feasibility and efficacy of BMC treatment in AMI patients. The patients enrolled in the study reach the 5 to 8 years FUP at 2011, raising the question whether the combined delivery of autologous BM-MNCs results in a long-term benefit for these patients.

Aim of the study: To investigate the long-term, 5 years clinical outcome of patients enrolled into the MYSTAR study.

Study design: Prospective non-randomized single-center Austrian long-term FUP registry.

Study patients: A total of 60 patients with previous cardiac stem cell therapy (participated in the MYSTAR study) will be included in the present study

Primary endpoint: occurrence of MACCE (major adverse cardiac and cerebrovascular events, including all-cause death, re-AMI, revascularization and stroke) during the mean 5 years follow-up.

Secondary endpoints: improvements of clinical symptoms, expressed as CCS and NYHA scores, change in global LV EF, measured by echocardiography, size of infarction determined by stress-rest SPECT, LV and RV volumes, function and cardiac output measured by cardiac MRI.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in the MYSTAR study, inclusion either in the Early or Late groups
* Signed informed consent

Exclusion Criteria:

* Non-willingness of participation in the present FUP study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included into the MYSTAR randomized study
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of MACCE | 5 years
  MACCE is defined as major adverse cardiac and cerebrovascular events including re-AMI, TVR, all-cause death and stroke at the 5-year FUP of the patients enrolled into the MYSTAR study and underwent cardiac stem cell therapy.

SECONDARY OUTCOMES:
Clinical symptoms (CCS, NYHA) | 5 years
Changes in global EF | 5 years
Size of infarction | 5 years
Left ventricular end-diastolic and end-systolic volumes | 5 years
Right ventricular end-diastolic and end-systolic volumes | 5 years
Right ventricular cardiac output | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mariann Gyöngyösi, MD PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Gyongyosi M, Giurgea GA, Syeda B, Charwat S, Marzluf B, Mascherbauer J, Jakab A, Zimba A, Sarkozy M, Pavo N, Sochor H, Graf S, Lang I, Maurer G, Bergler-Klein J; MYSTAR investigators. Long-Term Outcome of Combined (Percutaneous Intramyocardial and Intracoronary) Application of Autologous Bone Marrow Mononuclear Cells Post Myocardial Infarction: The 5-Year MYSTAR Study. PLoS One. 2016 Oct 20;11(10):e0164908. doi: 10.1371/journal.pone.0164908. eCollection 2016. PMID 27764157